CLINICAL TRIAL: NCT03011554
Title: A Prospective, Multicenter Clinical Trial of the Implantable Miniature Telescope in Pseudophakic Eyes With Central Vision Impairment Associated With End-Stage Macular Degeneration.
Brief Title: Telescope Exchange Study
Acronym: TES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IMT-TES-2016
Record Dates: First submitted 2017-01-02; First posted 2017-01-05 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Implantable Miniature Telescope (IMT) (Experimental): Intervention: Implanting the Implantable Miniature Telescope (IMT) in pseudophakic eyes of patients suffering from binocular end-stage AMD.
  Interventions: Device: Implantable Miniature Telescope (IMT)

INTERVENTIONS:
Device: Implantable Miniature Telescope (IMT) — Monocular implantation of the IMT.

SUMMARY:
VisionCare's Implantable Miniature Telescope (IMT, intraocular telescope or telescope) is indicated for monocular implantation to improve vision in eyes of patients at least 65 years of age with severe to profound vision impairment caused by bilateral central scotomas associated with end-stage age-related macular degeneration (AMD).

Patients with end-stage AMD who have undergone bilateral cataract removal and intraocular lens placement are currently contraindicated for telescope surgery.

These patients have no viable therapy available to improve their vision.

The objective of the TES pilot study is to evaluate the safety and effectiveness of implanting the intraocular telescope for improving vision in patients with bilateral end-stage age- related macular degeneration who are pseudophakic.

ELIGIBILITY:
Inclusion Criteria:

* Have retinal findings of geographic atrophy or disciform scar with foveal involvement as determined by FA
* Be age 65 or older
* Have BCDVA between 20/160 to 20/800 (inclusive) on ETDRS chart
* Be pseudophakic in the eye selected for telescope implantation
* Agree to undergo pre-surgery training with a low vision specialist
* Achieve at least a 5-letter improvement on the ETDRS chart with an external telescope
* Agree to participate in postoperative vision training with a low vision specialist.
* Patients must be able to provide and sign a voluntary informed consent.
* Patients must not meet any of the exclusion criteria below.

Exclusion Criteria:

* Stargardt's macular dystrophy
* Cognitive impairment that would interfere with the ability to understand instructions, follow directions, or prevent proper visual training/rehabilitation with the device.
* Any ophthalmic pathology that compromises fellow-eye peripheral vision
* A history of steroid-responsive rise in intraocular pressure (IOP), uncontrolled glaucoma, or preoperative IOP >22mmHg while on maximum medication
* Known sensitivity to planned study concomitant medications.
* An ocular condition that predisposes the patient to eye rubbing.
* Patients participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.
* Operative eye with:

  * Evidence of active CNV or treatment of CNV within 6 months
  * IOLs of the following types: PMMA, Crystalens, Tetraflex, Synchrony.
  * Central anterior chamber depth (ACD) < 3.0 mm; measurement of the ACD should be taken from the posterior surface of the cornea (endothelium) to the anterior surface of the IOL.
  * Axial length < 21 mm or >27 mm
  * Endothelial cell density (ECD) lower than 2300 cells/mm2 for subjects between the ages 65-69, lower than 2000 cells/mm2 for subjects between the ages of 70-74, and lower than 1800 cells/mm2 for subjects 75 years old or greater.
  * Corneal stromal or endothelial dystrophies, including guttata
  * History of intraocular or corneal surgery (including DSEK) except cataract removal and IOL placement
  * History of complicated cataract surgery
  * Compromised capsular bag (previous YAG posterior capsulotomy, evidence of tearing)
  * History of Radial Keratotomy
  * Inflammatory ocular disease
  * Pseudoexfoliation or zonular weakness
  * Diabetic retinopathy
  * Untreated retinal tears
  * Retinal vascular disease
  * Optic nerve disease
  * A history of retinal detachment
  * Intraocular tumor
  * Retinitis pigmentosa
  * Prior or expected ophthalmic related surgery within 30 days preceding telescope implantation
  * Any medical or ophthalmic condition that in the opinion of the investigator renders the subject unsuitable for participation in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Subjects will be followed up for three years post implantation
  All reported adverse events will be summarized by number and percent of occurence.

SECONDARY OUTCOMES:
Decrease in best corrected distance visual acuity (BCDVA) | Subjects will be followed up for three years post implantation
  Change in LogMar BCDVA from pre-operative visit will be summarized starting at 1 month post-op.
Endothelial Cell Density | Subjects will be followed up for three years post implantation
  ECD change and % change from preoperative visit will be summarized at each visit starting at 3 months post-op.

OTHER OUTCOMES:
Increase in best corrected distance visual acuity (BCDVA) | Subjects will be followed up for three years post implantation
  Change in LogMar BCDVA from pre-operative visit will be summarized starting at 1 month post-op.

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Garg, MD, Principal Investigator — University of California, Irvine; Derek Kunimoto, MD, Principal Investigator — Retinal Consultants of AZ
Locations (14):
- United States (14):
  - Retinal Consultants of AZ, Phoenix, Arizona
  - UC Irvine, Gavin Herbert Eye Institute, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Eye Physicians of Long Beach, Long Beach, California
  - Eye Care of San Diego, San Diego, California
  - Orange County Retina, Santa Ana, California
  - Sarasota Retina Institute, Sarasota, Florida
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Minnesota Eye Consultants, Minnetonka, Minnesota
  - Associated Eye Care, Stillwater, Minnesota
  - St. John's Clinic - Eye Specialists. Mercy, Springfield, Missouri
  - Eye Associates of New Mexico Vision Research Center, Albuquerque, New Mexico
  - Eye Specialty Group, Memphis, Tennessee
  - Cornea Consultants of Texas, Fort Worth, Texas